CLINICAL TRIAL: NCT05660408
Title: RNA PRIME - RNA Lipid Particles Targeting Pediatric Recurrent Intracranial Malignancies and Other systEmic Solid Tumors
Brief Title: RNA Lipid Particles Targeting Pediatric Recurrent Intracranial Malignancies and Other systEmic Solid Tumors
Acronym: RNA PRIME
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The V Foundation for Cancer Research (Other); National Pediatric Cancer Foundation (Other); Alex's Lemonade Stand Foundation (Industry); The Osteosarcoma Institute (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC23450; OCR43060 (Other: University of Florida); MCC23450 (Other: Moffitt Cancer Center)
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Pulmonary Osteosarcoma; Recurrent High-grade Glioma
Keywords: pulmonary osteosarcoma; RNA-LP; vaccines; immunotherapy; high-grade glioma; brain tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Recurrent pHGG, Arm 1 (Experimental): pHGG Arm 1-A single dose of pp65 RNA-LP (DP1) will be administered prior to standard of care surgical resection/biopsy, followed by at least two adjuvant DP1. During production of pp65/tumor mRNA RNA-LP (DP2) vaccines, treatment with DP1 will continue every 2 weeks. DP1 vaccines may continue until production of DP2 is complete (expected 5-8 weeks following initial surgery/biopsy).
  pp65/tumor mRNA RNA-LP (DP2) vaccinations will begin 7-14 days after the last dose of pp65 RNA-LP (DP1). DP2 treatment will occur approximately every 2 weeks for the first 3 doses. Following the first 3 doses of DP2, patients will receive 9 cycles of monthly DP2 for a total of 12 DP2 vaccines (minimum of 15 overall vaccines).
  Interventions: Biological: pp65 RNA LP (DP1); Biological: pp65/tumor mRNA RNA-LP (DP2); Procedure: Surgical Biopsy/Resection
- Recurrent pHGG, Arm 2 (Experimental): pHGG Arm 2-Standard of care surgical resection/biopsy will occur first and all three pp65 RNA-LP (DP1) will be administered in the adjuvant setting. During production of DP2, treatment will begin with DP1 every 2 weeks, beginning a minimum of 7-14 days after surgery/biopsy. DP1 vaccines may continue until production of DP2 is complete (expected 5-8 weeks following initial surgery/biopsy).
  pp65/tumor mRNA RNA-LP (DP2) vaccinations will begin 7-14 days after the last dose of pp65 RNA-LP (DP1). DP2 treatment will occur approximately every 2 weeks for the first 3 doses. Following the first 3 doses of DP2, patients will receive 9 cycles of monthly DP2 for a total of 12 DP2 vaccines (minimum of 15 overall vaccines).
  Interventions: Biological: pp65 RNA LP (DP1); Biological: pp65/tumor mRNA RNA-LP (DP2); Procedure: Surgical Biopsy/Resection
- Arm 1-Patients with unilateral pulmonary-only metastatic recurrent OSA (Experimental): OSA Arm 1-Patients with unilateral pulmonary-only metastatic recurrent OSA
  Participants will undergo surgical resection for sterile collection of tumor material to make pp65/tumor mRNA RNA-LP (DP2). During production of DP2 vaccines, participants will begin treatment with off-the-shelf pp65 RNA-LP (DP1) vaccines every 2 weeks. A minimum of 3 DP1 vaccines will be administered and may continue until production of DP2 is complete (expected 5-8 weeks following initial surgery/biopsy).
  DP2 vaccinations will begin 7-14 days after the last dose of DP1. DP2 treatment will occur approximately every 2 weeks for the first 3 doses. Participants will receive 9 cycles of monthly DP2 for a total of 12 DP2 vaccines (minimum of 15 overall vaccines).
  Interventions: Biological: pp65 RNA LP (DP1); Biological: pp65/tumor mRNA RNA-LP (DP2); Procedure: Surgical Biopsy/Resection
- Arm 2-Patients with bilateral pulmonary-only metastatic recurrent OSA (Experimental): OSA Arm 2-Patients with bilateral pulmonary-only metastatic recurrent OSA
  Participants will undergo surgical resection for sterile collection of tumor material to make pp65/tumor mRNA RNA-LP (DP2). For subjects in Arm 2, surgery will be again performed on contralateral lung nodules within 7 days following DP1 Vaccine #3.
  During production of pp65/tumor mRNA RNA-LP (DP2) vaccines, participants will begin treatment with off-the-shelf pp65 RNA-LP (DP1) vaccines every 2 weeks. A minimum of 3 DP1 vaccines will be administered and may continue until production of DP2 is complete (expected 5-8 weeks following initial surgery/biopsy). DP2 vaccinations will begin 14 days after 2nd surgical pulmonary metastectomy. DP2 treatment will occur approximately every 2 weeks for the first 3 doses. Participants will receive 9 cycles of monthly DP2 for a total of 12 DP2 vaccines (minimum of 15 overall vaccines).
  Interventions: Biological: pp65 RNA LP (DP1); Biological: pp65/tumor mRNA RNA-LP (DP2); Procedure: Surgical Biopsy/Resection
- Arm 3-Patients with unresectable OSA in any location (Experimental): Arm 3-Patients with unresectable OSA in any location.
  Participants will undergo surgical biopsy for sterile collection of tumor material to make pp65/tumor mRNA RNA-LP (DP2). For adult subjects only in Arm 3, optional biopsy will be repeated within 7 days following DP2 Vaccine #3 administration once hematologic recovery to eligibility criteria, unless medically contraindicated.
  During production of DP) vaccines, participants will begin treatment with off-the-shelf pp65 RNA-LP (DP1) vaccines every 2 weeks, beginning a minimum of 7 days after initial surgery/biopsy. A minimum of 3 DP1 vaccines will be administered and may continue until production of DP2 is complete (expected 5-8 weeks following initial surgery/biopsy). DP2 vaccinations will begin 7-14 days after the last dose of DP1. DP2 treatment will occur approximately every 2 weeks for the first 3 doses. Participants will receive 9 cycles of monthly DP2 for a total of 12 DP2 vaccines (minimum of 15 overall vaccines).
  Interventions: Biological: pp65 RNA LP (DP1); Biological: pp65/tumor mRNA RNA-LP (DP2); Procedure: Surgical Biopsy/Resection

INTERVENTIONS:
Biological: pp65 RNA LP (DP1) — This is an off the shelf RNA-LP vaccine used to prime for the immune response while we produce the patient specific pp65/tumor mRNA RNA-LP (DP2)
Biological: pp65/tumor mRNA RNA-LP (DP2) — This is a patient specific RNA-LP vaccine generated from the patient's tumor RNA.
Procedure: Surgical Biopsy/Resection — Eligible participants will be enrolled and undergo sterile collection of tumor material .

SUMMARY:
The Investigators have demonstrated in preclinical studies that RNA liposomes activate APCs, induce antigen-specific T cell immunity, and can supplant DCs in a cell therapy model for HGG and have shown feasibility and activity of this approach in preclinical models and in canine patients with a spontaneous malignant glioma. In one arm of this study, we will investigate the safety and immunologic activity of RNA-LP vaccines in pediatric patients with recurrent pHGG.

The investigators have also shown that intravenous administration of tumor mRNA loaded lipid particles (LPs) localizes primarily to lung, transfect antigen presenting cells (APCs) and lead to an activated T cell response for induction of anti-tumor immunity. In contrast to other formulations, RNA-LPs recruit multiple arms of the immune system (i.e. innate/adaptive), and remodel the systemic/intratumoral immune milieu, which remain potent barriers for vaccine, cellular, and checkpoint inhibiting immunotherapies. After only a single RNA-LP vaccine, the bulk of systemic and intratumoral dendritic cells (DCs) in mice display an activated phenotype; these activated DCs (harvested from tumors) expand antigen specific T cell immunity. In immunologically resistant pulmonary osteosacroma murine tumor models (i.e. K7M2), RNA-LPs induce robust anti-tumor efficacy in settings where immune checkpoint inhibitors (i.e. anti-PD-L1 therapy) do not confer therapeutic benefit. The investigators have already demonstrated safety of RNA-LPs in acute/chronic murine toxicity studies, and in client-owned canine trial.

In this study, we will investigate the manufacturing feasibility, safety and immunologic activity of RNA-LP vaccine in patients with recurrent pulmonary or unresectable osteosarcoma and recurrent pHGG.

DETAILED DESCRIPTION:
For recurrent pHGG there will be two non-randomized arms assigned at the discretion of the patient and treatment team:

* Arm 1-A single neoadjuvant pp65 RNA-LP (DP1) will be administered prior to surgical resection/biopsy, and then two adjuvant DP1.
* Arm 2-Surgical resection/biopsy will occur first and all three DP1 will be administered in the adjuvant setting

For recurrent OSA there will be three arms based on disease status on enrollment:

* Arm 1-Patients with unilateral pulmonary-only metastatic recurrent OSA
* Arm 2-Patients with bilateral pulmonary-only metastatic recurrent OSA
* Arm 3-Patients with unresectable OSA in any location.

The Phase I dose-escalation study for either recurrent/progressive pHGG or recurrent OSA cohort will be performed in 18 subjects using a 3+3 design. Both recurrent pHGG trial arms will be enrolled together as a single cohort for safety, and similarly all recurrent OSA trial arms will be enrolled together as a single cohort for safety during phase I.

ELIGIBILITY:
Inclusion Criteria:

Patients with recurrent or progressive pediatric high-grade glioma (pHGG)

Patients must be age 3-25 years

Diagnosis:

Patients must have had a prior histologically-diagnosed pHGG(including but not limited to: Astrocytoma WHO Grade 3 or 4 and Glioblastoma WHO Grade 4 by histopathology or molecular studies, per 2021 WHO Classification of Tumors of the CNS57, WHO CNS5).

* Patients with M+ disease without gliomatosis cerebri (see definition under exclusion criteria) ARE eligible.
* Recurrent pHGG involving the midline structures other than those intrinsically located within the pons ARE eligible.
* Patients with mismatch repair deficient (MMRD) tumors refractory to immune checkpoint inhibitors ARE eligible.

Patients must have recurred or progressed after receiving surgery/biopsy and radiation therapy as frontline standard-of-care treatments in primary disease.

Patients must have MRI evidence of probable recurrent pHGG. Patients must be clinically eligible for standard-of-care surgical resection/biopsy and sterile collection of tumor material in a manner suitable for RNA extraction, amplification, and loading of lipid particles.

Performance Level Karnofsky ≥ 60% for patients ≥ 16 years of age and Lansky ≥ 60% for patients ≤ 16 years of age

* Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participants with post-surgical neurological deficits should have deficits that are stable for a minimum of 2 week prior to enrollment.

Prior Therapy

Patients must have recovered from all acute toxic effects of all prior anti-cancer therapy (all adverse events must have improved to grade 1 or better):

* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: ≥ 21 days after the last dose of myelosuppressive chemotherapy. If questions, the agent and duration can be discussed with the study chair.
* Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or ANC counts): ≥ 14 days after the last dose of agent. If questions, the agent and duration can be discussed with the study chair.
* Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
* Corticosteroids: All systemically administered corticosteroids must be stable or decreasing for ≥ 1 week prior to enrollment, with a maximum dexamethasone dose of 2.8 mg/m2/day. Corticosteroid physiologic replacement therapy for management of pituitary/adrenal axis insufficiency and/or topical administration (e.g. inhaled or dermatologic) is allowed.
* Hematopoietic growth factors: ≥14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or ≥7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Interleukins, Interferons, and Cytokines (other than hematopoietic growth factors): ≥ 21 days after the completion of interleukins, interferon, or cytokines.
* Stem cell infusions (with or without TBI):

  * Autologous stem cell infusion including boost infusion: ≥ 30 days.
* Cellular Therapy: ≥ 42 days after the completion of any type of cellular therapy (e.g., modified T cells, NK cells, dendritic cells, etc.)
* XRT/External Beam Irradiation, including Protons: ≥ 90 days after local XRT unless recurrence is a new enhancement on MRI outside the radiation treatment field; ≥ 150 days after TBI, craniospinal XRT or if radiation to ≥ 50% of the pelvis.
* Radiopharmaceutical therapy (e.g., radiolabeled antibody): ≥ 42 days after systematically administered radiopharmaceutical therapy.
* Other therapeutic clinical trials: ≥ 14 days after last dose of investigational agent, unless otherwise defined above.
* Prior use of RNA-LP therapy: Patients must not have received prior exposure to pp65-directed therapy or any RNA-LP therapy.

Organ Function Requirements

Adequate bone marrow function as defined as:

* Absolute neutrophil count (ANC) ≥ 1,000/µl
* Platelets ≥ 100,000/µl (transfusion-independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin ≥ 8 g/dL (transfusion-independent, defined as not receiving packed red blood cell transfusions for at least 7 days prior to enrollment)

Adequate renal function as defined as:

* A creatinine based on age/gender
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2

Adequate liver function as defined as:

* Total bilirubin ≤ 3x institutional upper limits of normal for age
* ALT ≤ 5x institutional upper limits of normal for age
* AST ≤ 5x institutional upper limits of normal for age Adequate pulmonary function defined as baseline pulse oximetry of at least 92% on room air.

All patients must be willing to take an antiepileptic medication such as levetiracetam for the duration of RNA-LP vaccinations.

Contraception

* Women of childbearing potential must agree to use of at least 2 forms of acceptable contraceptive methods or abstinence to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.
* Men with female partners of childbearing potential must agree to use of at least 2 forms of acceptable contraceptive methods or abstinence throughout the study and should avoid conceiving children for at least 24 weeks following the last dose of study drug.

All patients and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent/assent document.

Inclusion Criteria:

Patients with osteosarcoma (OSA)

Age: Patients must be age 3-39 years. Diagnosis

* For Arms 1 and 2: Patients must be clinically eligible for standard-of-care surgical resection of suspected OSA recurrence with pulmonary-only metastases.
* For Arm 3: Patients must undergo standard-of-care biopsy of suspected or known recurrent, unresectable OSA.

Disease Status

* For Arm 1: Patients must be eligible for single-sided thoracotomy for planned surgical resection of all OSA pulmonary metastases.
* For Arm 2: Patients must be eligible for staged two-sided thoracotomies for planned surgical resection of all OSA pulmonary metastases.
* For Arm 3: Patients must have unresectable OSA. Patients must have sufficient disease on diagnostic contrast-enhanced MRI wherein surgical biopsy is feasible.

Patients must have sterile collection of tumor material in a manner suitable for RNA extraction, amplification, and loading of lipid particles.

Performance Level: Karnofsky ≥ 60% for patients > 16 years of age and Lansky ≥ 60% for patients < 16 years of age.

* NOTE: Participants who are unable to walk because of amputation, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior Therapy: Patients must have recovered from all acute toxic effects of all prior anti-cancer therapy (all adverse events must have improved to grade 1 or better):

Prior Therapy: Patients must have recovered from all acute toxic effects of all prior anti-cancer therapy (all adverse events must have improved to grade 1 or better):

1. Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: ≥ 14 days after the last dose of myelosuppressive chemotherapy. If questions, the agent and duration can be discussed with the study chair.
2. Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or ANC counts): ≥ 7 days after the last dose of agent. If questions, the agent and duration can be discussed with the study chair.
3. Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
4. Corticosteroids: All systemically administered corticosteroids must be stable or decreasing for ≥ 1 week prior to enrollment, with a maximum dexamethasone dose of 2.8 mg/m2/day. Corticosteroid physiologic replacement therapy for management of pituitary/adrenal axis insufficiency and/or topical administration (e.g. inhaled or dermatologic) is allowed.
5. Hematopoietic growth factors: ≥ 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or ≥ 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
6. Interleukins, Interferons, and Cytokines (other than hematopoietic growth factors): ≥ 21 days after the completion of interleukins, interferon, or cytokines.
7. Stem cell infusions (with or without TBI): Autologous stem cell infusion including boost infusion: ≥ 30 days.
8. Cellular Therapy: ≥ 42 days after the completion of any type of cellular therapy (e.g., modified T cells, NK cells, dendritic cells, etc.).
9. XRT/External Beam Irradiation, including Protons: ≥ 90 days after local XRT unless recurrence is a new enhancement on MRI outside the radiation treatment field; ≥ 150 days after TBI or if radiation to ≥ 50% of the pelvis; ≥ 42 days if other substantial BM radiation.
10. Radiopharmaceutical therapy (e.g., radiolabeled antibody): ≥ 42 days after systematically administered radiopharmaceutical therapy.
11. Other therapeutic clinical trials: ≥ 14 days after last dose of investigational agent, unless otherwise defined above
12. Prior use of RNA-LP therapy: Patients must not have received prior exposure to pp65-directed therapy or any RNA-LP therapy.

Organ Function Requirements

Adequate bone marrow function as defined as:

* Absolute neutrophil count (ANC) ≥ 1,000/µl
* Platelets ≥ 100,000/µl (transfusion-independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin ≥ 8 g/dL (transfusion-independent, defined as not receiving packed red blood cell transfusions for at least 7 days prior to enrollment)

Adequate renal function as defined as:

* A creatinine based on age/gender
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2

Adequate liver function as defined as:

* Total bilirubin ≤ 3x institutional upper limits of normal for age
* ALT ≤ 5x institutional upper limits of normal for age
* AST ≤ 5x institutional upper limits of normal for age Adequate pulmonary function defined as baseline pulse oximetry of at least 92% on room air.

Contraception

* Women of childbearing potential must agree to use of at least 2 forms of acceptable contraceptive methods or abstinence to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.
* Men with female partners of childbearing potential must agree to use of at least 2 forms of acceptable contraceptive methods or abstinence throughout the study and should avoid conceiving children for at least 24 weeks following the last dose of study drug.

All patients and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent/assent document.

Exclusion Criteria for all Strata

Diagnosis

* Diffuse intrinsic pontine glioma
* Gliomatosis cerebri - clear tumor involvement of multiple areas (>3 lobes), OR presence of clinical and/or radiographic evidence of impending herniation or spinal cord compression.

NOTE: review by Study Chairs is recommended

Patients who are receiving any other investigational agents.

Pregnancy or Breastfeeding

o Pregnant or breastfeeding women will not be entered on this study because there is no available information regarding human fetal or teratogenic toxicities. Females of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to starting protocol therapy.

Severe, active co-morbidity, including, but not limited to:

* Known active immunosuppressive disease.
* Unstable angina and/or congestive heart failure requiring hospitalization.
* Unstable cardiac arrhythmias, abnormalities, or transmural myocardial infarction within the last 6 months.
* Uncontrolled infection
* Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other known respiratory illness requiring hospitalization or precluding study therapy
* Hepatic insufficiency resulting in clinical jaundice and/or clinically significant coagulation defects.
* Patients with autoimmune disease requiring medical management with immunosuppressants.
* Prior history of brachial neuritis or Guillain-Barre syndrome.
* Uncontrolled seizure disorder
* Major medical illnesses or psychiatric impairments that, in the investigators' opinions, will prevent administration or completion of protocol therapy.

History of myocarditis

Receipt of any live vaccine within 30 days prior to day 1 of treatment.

Patients who have received an allogeneic (non-autologous) bone marrow or stem cell transplant, or any allogeneic stem cell infusion including DLI or boost infusion.

Participants who are unwilling or unable to receive treatment and undergo follow-up evaluations, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 14 months
  Determine the maximum tolerated dose of RNA-LP vaccine based on frequency of dose-limiting toxicities.
Feasibility of generating RNA-LP | 14 months
  Ability to generate patient-specific pp65/tumor mRNA RNA-LP that meet release criteria.

SECONDARY OUTCOMES:
Overall survival rate | 3 years
  Determine the survival in patients with recurrent pHGG or oseteosarcoma receiving RNA-LP vaccine.
Immune activation | 3 years
  Determine if immune cells in patients receiving RNA-LPs become activated in both peripheral blood and in the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: John Ligon, MD, Study Chair — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

REFERENCES:
- [Derived] Villanueva MT. RNA delivery heats up cold tumours. Nat Rev Drug Discov. 2024 Jul;23(7):497. doi: 10.1038/d41573-024-00098-0. No abstract available. PMID 38858569